CLINICAL TRIAL: NCT03762330
Title: Effect of a Structured Comprehensive Intervention to Stimulate Self- Management and Improve Quality of Life in People With Chronic Obstructive Pulmonary Disease(COPD). A Randomised Clinical Trial.
Brief Title: Structured Comprehensive Intervention to Stimulate Self- Management and Improve Quality of Life in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Catala de Salut (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P17/055
Record Dates: First submitted 2018-11-14; First posted 2018-12-03 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: quality of life; self-management,; structured plan; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD structured self-management plan (Active Comparator): Participants will receive usual care for COPD and in addition, a structured self-management education plan.
  Interventions: Behavioral: COPD structured self-management plan.
- Usual care (No Intervention): COPD participants receiving only usual care

INTERVENTIONS:
Behavioral: COPD structured self-management plan. — Education plan , including knowledge of the disease, healthy life habits, correct use of inhalers, skills to control symptoms and strategies to face the disease and exacerbations
  Arms: COPD structured self-management plan

SUMMARY:
This study evaluates the effect of of a structured self-management intervention plan in patients with chronic obstructive pulmonary disease in primary care setting.Half of the participants will receive the self-management plan while the other half will receive usual care.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a great magnitude public health problem with an associated increased mortality and a high cost (consumption of health care resources and loss of health related quality of life (HRQoL)). The comprehensive approach to this complex disease, focusing self-care promotion, improves HRQoL and the patients" clinical status, as shown by several studies, although further investigation is needed to confirm these results in the field of Primary Care (PC) and to formulate clear recommendations on the more effective type of intervention.

Hypothesis: In (moderate-severe) COPD patients, a structured self-management intervention plan in the setting of primary care, is more effective than usual treatment on the main outcomes associated with the disease: HRQoL, lung function, exacerbations and hospital admissions, at 6, 12 and 24 months of follow-up.

Objectives: To evaluate the impact of a comprehensive intervention plan to promote self-care and improve HRQoL in people with COPD in PC.

Methods: Multicenter randomized controlled trial, conducted at PC centers in Barcelona.

Determinations: Specific standardized and validated questionnaires, as the St George's Respiratory for the HRQoL. Statistical analysis: Intention to treat analysis. Descriptive statistics of the variables of the intervention and the control group to assess their homogeneity at the beginning of the study. An analysis of variance (ANOVA) will be used to assess differences among intervention groups.

Expected results: A significant improvement in HRQoL attributable to the intervention performed in patients with COPD Applicability and Relevance: To implement the intervention plan in clinical practice and to standardize its content.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one visit at the primary care physician during the past year
* Patients with a diagnosis of moderate (FEV1 50% - 80%) or severe (FEV1 30% - 50%) COPD
* Patients treated with inhaled bronchodilators and accepting to participate in the study.

Exclusion Criteria:

* Patients unable to come to the primary care centre
* Patients with cognitive impairment and/or a severe mental condition.
* Patients with a diagnosis of asthma, tuberculosis or other chronic respiratory disease.
* Patients needing chronic oxygen therapy.
* Patients with any terminal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-19 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life St. George´s Respiratory Questionnaire (SGRQ) | Change from baseline at 6 ,12 and 24 months
  St. George´s Respiratory Questionnaire (SGRQ).Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.
  Number of items: 50 items Number of domains & categories : 2 parts (3 components). Part 1 : Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall.
  Scaling of items Part I (Symptoms): several scales; Part II (Activity and Impacts): dichotomous (true/false) except last question (4-point Likert scale). Scores range from 0 to 100, with higher scores indicating more limitations.

SECONDARY OUTCOMES:
Intensity of symptoms related to COPD | Change from baseline at 6 ,12 and 24 months
  COPD Assessment Test (CAT) : It consists of 8 questions with 5 possible answers valued from 0 to 5 (values close to 0: better health status)
Dyspnea score severity | Change from baseline at 6 ,12 and 24 months
  Dyspnea severity assessed by the modified scale of the Medical Research Council (mMRC). Range 0-4 (none to maximum)
Changes in the Body mass index, Obstruction, Dyspnea, Exacerbations Index (BODEx index ) | Change from baseline at 6 ,12 and 24 months
  Index including BMI (Body mass index), Obstruction, Dyspnea, Exacerbations. with possible answers from 0-3, each item. Range: 0-9. Mild: 0-2 Moderate: 3-4 Severe ≥5
Number of COPD exacerbations | at 6 ,12 and 24 months from baseline
  Number of COPD exacerbations requiring a visit to primary care physician
Number of hospital admissions due to COPD exacerbation | at 6 ,12 and 24 months from baseline
  Number of hospital admissions due to COPD exacerbation
Changes in Anxiety and depression scales | Change from baseline at 6 ,12 and 24 months
  Goldberg's anxiety-depression scale (GADS): is an 18-item self-report symptom inventory that was developed by Goldberg and colleagues from 36 items in the Psychiatric Assessment Schedule. The GADS score is based on responses of 'yes' or 'no' to nine depression and nine anxiety items, asking how respondents have been feeling in the past month. Goldberg et al. (1988) considered patients with anxiety scores of 5 or more or with depression scores of 2 or more as having a 50% chance of a clinically important disturbance
Changes in forced vital capacity (FVC) | Change from baseline at 6 ,12 and 24 months
  Value of FVC measured with forced spirometry
Changes in forced expiratory volume at the first second (FEV1) | Change from baseline at 6 ,12 and 24 months
  Value of FEV1 measured with forced spirometry
Results of the Test of Adherence to Inhalers (TAI test) | Change from baseline at 6 ,12 and 24 months
  TAI test. Includes 10 questions self-completed by patient. Range of each questions; 1worse compliance and 5 best compliance. The total score of the 10 items gives a total from 1-50.
Use of long-acting beta-adrenergic bronchodilator in monotherapy | At baseline and at 6 ,12 and 24 months
  Use of long-acting beta-adrenergic bronchodilator in monotherapy (yes or no)
Use of long-acting anticholinergic bronchodilator in monotherapy | At baseline and at 6 ,12 and 24 months
  Use of long-acting anticholinergic bronchodilator in monotherapy (yes or no)
Use of a double therapy of long-acting beta-adrenergic bronchodilator and long-acting anticholinergic bronchodilator | At baseline and at 6 ,12 and 24 months
  Use of a double therapy of long-acting beta-adrenergic bronchodilator and long-acting anticholinergic bronchodilator (yes or no)
Use of a double therapy of long-acting beta-adrenergic bronchodilator and short-acting anticholinergic bronchodilator | At baseline and at 6 ,12 and 24 months
  Use of a double therapy of long-acting beta-adrenergic bronchodilator and short-acting anticholinergic bronchodilator (yes or no)
Use of a triple therapy of long-acting beta-adrenergic bronchodilator and long-acting anticholinergic bronchodilator plus inhaled steroids | At baseline and at 6 ,12 and 24 months
  Use of a triple therapy of long-acting beta-adrenergic bronchodilator plus long-acting anticholinergic bronchodilator plus inhaled steroids (yes or no)
Use of a triple therapy of long-acting beta-adrenergic bronchodilator and short-acting anticholinergic bronchodilator plus inhaled steroids | At baseline and at 6 ,12 and 24 months
  Use of a triple therapy of long-acting beta-adrenergic bronchodilator and short-acting anticholinergic bronchodilator plus inhaled steroids (yes or no)
Use of Roflumilast | At baseline and at 6 ,12 and 24 months
  Use of Roflumilast (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Maite Lopez Luque, Principal Investigator — Servei Catala de la Salut
Locations (1):
- EAP Montcada i Reixac, Barcelona, Spain

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT03762330/Prot_SAP_000.pdf